CLINICAL TRIAL: NCT04545996
Title: Effects of Sub-Occipital Muscles Inhibition Technique and Cranio Cervical Flexion Exercise for Mechanical Neck Pain
Brief Title: Sub-Occipital Muscles Inhibition Technique Verses Cranio Cervical Flexion Exercise for Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00682 Robina Malik
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Cervical Pain; Mechanical Neck Pain
Keywords: Sub-Occipital Muscles Inhibition Technique; Cranio Cervical Flexion Exercise
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Rang of Motion Exercises. (Active Comparator): Cervical exercises for mechanical neck pain.
  Interventions: Other: Suboccipital Inhibition Technique
- Cervical Exercises. (Experimental): Cervical exercises for the management of mechanical neck pain.
  Interventions: Other: Cranio Cervical Flexion Exercises.

INTERVENTIONS:
Other: Suboccipital Inhibition Technique — Suboccipital Inhibition Technique For 2min And Conventional Treatment Hot Pack For 10 To 15 Mints And Muscle Energy Technique(Post Facilitation Stretch) 5 Reps × 1 Set Sessions: 2 TIME A WEEK FOR 4 CONSECUTIVE WEEKS
  Arms: Cervical Rang of Motion Exercises.
Other: Cranio Cervical Flexion Exercises. — Cranio cervical flexion exercises10 repetitions for 10 seconds and conventional treatment hot pack for 10 to 15 mints and muscle energy technique(post facilitation stretch) 5 reps × 1 set Sessions: 2 TIME A WEEK FOR 4 CONSECUTIVE WEEKS
  Arms: Cervical Exercises.

SUMMARY:
The aim of this research is to determine the Effects of Sub-Occipital Muscles Inhibition Technique and Cranio Cervical Flexion Exercise for Mechanical Neck Pain. A randomized control trail will conduct at Railway general hospital(IIMCT). The sample size will be 68. TheParticipants will bedividing into two groups,34 participants in Group A (receive the Sub-Occipital Muscles Inhibition Technique) and 34 in Group B (receive Cranio Cervical Flexion Exercise). The study duration will 6 months. Purposive non probability sampling technique will be applied. Both male and female participants with mechanical neck pain will be include. Tools use in this study areNumerical Pain Rating Scale (NPRS), Neck Disability Index (NDI),Goniometer, Pressure Biofeedback unit, Digital Camera. Data analyzed through SPSS version 21.

DETAILED DESCRIPTION:
Mechanical neck pain (MNP) is generalized neck or shoulder pain with mechanical characteristics (including symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature). It has become an increasing problem causing functional disability in large populations. It is one of the most common musculoskeletal disorders in the neck region. Neck pain of mechanical origin constitutes approximately 45% - 50% of all neck pain. The variation in the prevalence ranges from 43.0% of the Swedish population, 34.4% of Norwegian adult population and In North America (Saskatchewan, Canada) lifetime prevalence of neck pain is 66.7%. The reason for this may lie in the increasing time spent on office and computer work. Also, a significant proportion of mechanical neck disorders consist of whiplash associated disorders (WAD), with a higher prevalence in women (22%) than in men (16%). Strong evidence suggests biomechanical factors, including prolonged computer use, and posture and repetitive movements are associated with the development of neck pain. Cervical joint dysfunction is the main cause of mechanical neck pain. One of the predominant mechanical events causing neck pain, is impaired stability of the cervical spine, which is often attributed to disturbances in motor control over the cervical spine. The stability of the cervical spine is dependent on the deep neck flexor and neck extensor muscles. The longuscolli and capitis are principal deep neck flexor muscles. In contrast, the suboccipital muscles are principal neck extensors of the upper cervical spine and are composed of the rectus capitis posterior major (RCPM), rectus capitis posterior minor (RCPm), obliquuscapitis superior (OCS), and obliquuscapitis inferior (OCI). There are varieties of physiotherapy interventions for the management of Mechanical neck pain such as spinal joint manipulation, mobilization techniques, massage techniques, suboccipital muscle inhibition technique, craniocervical flexion exercise, soft tissue techniques and trigger point [TrP] treatment , needling, active release techniques, stretches (static and isometric ), traction and various electro modalities.A very limited evidence found on comparison on effectiveness of sub occipital muscle release and Cranio-cervical flexion exercise. Previous studies only find out immediate effect (one session) on Cervical ROM and CVA. To fill the gap, this study is formulated to determine the effects of sub occipital muscle release and Cranio-cervical flexion exercise on ROM in the cervical spine and Cranio-vertebral angle (CVA) in mechanical neck pain. Study will find out most effective treatment for management of mechanical neck pain and would contribute to educate and treat the patient with most simple and effective treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* At least five points on the neck disability index (NDI)
* 3 to 6 points in the numerical pain rating scale (NPRS)
* pain from more than 3 months
* Subjects were included if they had FHP as determined by the presence of a CVA < 48
* Subjects will include if they have flexion <80°, extension<70°, lateral flexion <20° and rotation <90

Exclusion Criteria:

* History of traffic accidents
* History of lower extremity fracture and surgery
* Acute low back and neck pain
* History of lumbar and cervical herniated intervertebral disk and spinal stenosis
* History of cervical spine surgery and trauma
* History of vascular disease in the head and neck
* Progressive neuro logical deficits

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 4th day.
  Changes from base line Northwick disability index was developed first in Northwick Park hospital, England. It was designed to measure the neck pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100.

SECONDARY OUTCOMES:
Numeric Pain Rating scale. | 4th day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain.
Cranio vertebral angle | 4th day
  Changes from the Baseline Cranio vertebral angle will taken with the help of digital camera.
Rang of Motion of cervical spine. | 4th day
  Changes from the Baseline range of Motion of cervical spine willtake with the Help of Goniometer.
Cervical flexion exercise. | 4th day
  Changes from the Baseline cervical flexion exercise will access by pressure biofeedback unit.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Iglesias J, Fernandez-de-las-Penas C, Cleland JA, Alburquerque-Sendin F, Palomeque-del-Cerro L, Mendez-Sanchez R. Inclusion of thoracic spine thrust manipulation into an electro-therapy/thermal program for the management of patients with acute mechanical neck pain: a randomized clinical trial. Man Ther. 2009 Jun;14(3):306-13. doi: 10.1016/j.math.2008.04.006. Epub 2008 Aug 8. PMID 18692428
- [Background] Celenay ST, Kaya DO, Akbayrak T. Cervical and scapulothoracic stabilization exercises with and without connective tissue massage for chronic mechanical neck pain: A prospective, randomised controlled trial. Man Ther. 2016 Feb;21:144-50. doi: 10.1016/j.math.2015.07.003. Epub 2015 Jul 15. PMID 26211422
- [Background] Jeong ED, Kim CY, Kim SM, Lee SJ, Kim HD. Short-term effects of the suboccipital muscle inhibition technique and cranio-cervical flexion exercise on hamstring flexibility, cranio-vertebral angle, and range of motion of the cervical spine in subjects with neck pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2018;31(6):1025-1034. doi: 10.3233/BMR-171016. PMID 30248030
- [Background] Guez M, Hildingsson C, Nilsson M, Toolanen G. The prevalence of neck pain: a population-based study from northern Sweden. Acta Orthop Scand. 2002 Aug;73(4):455-9. doi: 10.1080/00016470216329. PMID 12358121
- [Background] Bovim G, Schrader H, Sand T. Neck pain in the general population. Spine (Phila Pa 1976). 1994 Jun 15;19(12):1307-9. doi: 10.1097/00007632-199406000-00001. PMID 8066508
- [Background] Camitsis A. The effect of craniocervical flexion exercise on cervical posture and cervical range of motion in asymptomatic participants.
- [Background] Sarig-Bahat H. Evidence for exercise therapy in mechanical neck disorders. Man Ther. 2003 Feb;8(1):10-20. doi: 10.1054/math.2002.0480. PMID 12586557
- [Background] Lluch E, Arguisuelas MD, Coloma PS, Palma F, Rey A, Falla D. Effects of deep cervical flexor training on pressure pain thresholds over myofascial trigger points in patients with chronic neck pain. J Manipulative Physiol Ther. 2013 Nov-Dec;36(9):604-11. doi: 10.1016/j.jmpt.2013.08.004. Epub 2013 Oct 21. PMID 24152997
- [Background] Cleland JA, Childs JD, McRae M, Palmer JA, Stowell T. Immediate effects of thoracic manipulation in patients with neck pain: a randomized clinical trial. Man Ther. 2005 May;10(2):127-35. doi: 10.1016/j.math.2004.08.005. PMID 15922233
- [Background] Mejuto-Vazquez MJ, Salom-Moreno J, Ortega-Santiago R, Truyols-Dominguez S, Fernandez-de-Las-Penas C. Short-term changes in neck pain, widespread pressure pain sensitivity, and cervical range of motion after the application of trigger point dry needling in patients with acute mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):252-60. doi: 10.2519/jospt.2014.5108. Epub 2014 Feb 25. PMID 24568260
- [Background] Kim BB, Lee JH, Jeong HJ, Cynn HS. Effects of suboccipital release with craniocervical flexion exercise on craniocervical alignment and extrinsic cervical muscle activity in subjects with forward head posture. J Electromyogr Kinesiol. 2016 Oct;30:31-7. doi: 10.1016/j.jelekin.2016.05.007. Epub 2016 May 24. PMID 27261928
- [Background] Gonzalez Rueda V, Lopez de Celis C, Barra Lopez ME, Carrasco Uribarren A, Castillo Tomas S, Hidalgo Garcia C. Effectiveness of a specific manual approach to the suboccipital region in patients with chronic mechanical neck pain and rotation deficit in the upper cervical spine: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Sep 5;18(1):384. doi: 10.1186/s12891-017-1744-5. PMID 28870191
- [Background] Park SK, Yang DJ, Kim JH, Kang DH, Park SH, Yoon JH. Effects of cervical stretching and cranio-cervical flexion exercises on cervical muscle characteristics and posture of patients with cervicogenic headache. J Phys Ther Sci. 2017 Oct;29(10):1836-1840. doi: 10.1589/jpts.29.1836. Epub 2017 Oct 21. PMID 29184301
- [Background] Falla D, Jull G, Russell T, Vicenzino B, Hodges P. Effect of neck exercise on sitting posture in patients with chronic neck pain. Phys Ther. 2007 Apr;87(4):408-17. doi: 10.2522/ptj.20060009. Epub 2007 Mar 6. PMID 17341512
- [Background] Swartz EE, Floyd RT, Cendoma M. Cervical spine functional anatomy and the biomechanics of injury due to compressive loading. J Athl Train. 2005 Jul-Sep;40(3):155-61. PMID 16284634
- [Background] Shaghayegh Fard B, Ahmadi A, Maroufi N, Sarrafzadeh J. Evaluation of forward head posture in sitting and standing positions. Eur Spine J. 2016 Nov;25(11):3577-3582. doi: 10.1007/s00586-015-4254-x. Epub 2015 Oct 17. PMID 26476717